CLINICAL TRIAL: NCT00283608
Title: Pharmacogenetics of Aromatase Inhibitors
Brief Title: Pharmacogenetics of Anastrozole in Postmenopausal Women With Estrogen Receptor-Positive and/or Progesterone Receptor-Positive Stage I, Stage II, or Stage III Breast Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James N. Ingle, M.D., Mayo Clinic Cancer Center
Other Study IDs: CDR0000583001; MC0532 (Other: Mayo Clinic Cancer Center); 999-05 (Other: Mayo Clinic IRB); NCT00366054 (obsolete NCT alias)
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Polymorphism, Single Nucleotide; Chromatography, High Pressure Liquid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Anastrozole treatment group samples will be used as described for this study, and then will be destroyed.
  Exemestane treatment group samples of blood will be stored at Mayo Clinic Rochester.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Anastrozole: Blood draws for baseline and six to twelve weeks.
  Interventions: Genetic: Single nucleotide polymorphism (SNP); Other: high performance liquid chromatography; Other: measurements by DXA; Other: questionnaire administration
- Exemestane: Blood draws for baseline and six to twelve weeks
  Interventions: Genetic: Single nucleotide polymorphism (SNP); Other: high performance liquid chromatography; Other: measurements by DXA; Other: questionnaire administration

INTERVENTIONS:
Genetic: Single nucleotide polymorphism (SNP) — Evaluating SNP association with traits.
Other: high performance liquid chromatography — analysis of plasma concentrations of drugs
Other: measurements by DXA — determine bone mineral density (BMD)
Other: questionnaire administration — determine attitude changes

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients with cancer receiving anastrozole may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors learn more about how anastrozole works in the body.

PURPOSE: This research study is looking at the pharmacogenetics of anastrozole in postmenopausal women with estrogen receptor-positive (ER+) and/or progesterone receptor-positive (PR+) stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the association of intragenic haplotypes in genes encoding proteins involved in anastrozole metabolism pathways with anastrozole steady state plasma levels in postmenopausal women with estrogen receptor-positive and/or progesterone receptor-positive stage I, II, or III breast cancer.
* To evaluate the association of intragenic haplotypes in genes that encode proteins involved in pathways for estrogen synthesis, metabolism, and transport and in genes involved in anastrozole metabolism with the pharmacodynamic (PD) effects of anastrozole therapy, as measured by changes (before vs after drug therapy) in plasma levels of estradiol, estrone, estrone sulfate, testosterone, and androstenedione in these patients.
* To evaluate the association of intragenic haplotypes described above with the PD effects of anastrozole therapy, as measured by changes in breast density and bone mineral density before and at 1 year after drug therapy.
* To collect and bank blood samples and mammographic, bone density, and questionnaire data from patients enrolled on CAN-NCIC-MA27 and randomized to receive exemestane.

OUTLINE: This is a multicenter study. Patients are stratified according to prior tamoxifen use (yes vs no).

Blood samples are obtained for pharmacogenetic studies at baseline, at 6-12 weeks, and then at 1 year. Samples are analyzed for plasma anastrozole concentrations via high-performance liquid chromatography; genotyping for htSNPs via PCR; plasma levels of estradiol, estrone, estrone sulfate, testosterone, and androstenedione via gas chromatographic negative chemical ionization tandem mass spectrometry and liquid chromatographic electrospray tandem mass spectrometry.

Mammograms are obtained at baseline (i.e., within the past 6 months) and at 1 year to assess breast density. Patients with bilateral disease, bilateral breast augmentation, or bilateral mastectomy do not participate in this portion of the study.

Patients at the Mayo Clinic Cancer Center Rochester site also undergo bone mineral density measurement via dual x-ray absorptiometry at baseline and at 1 year. Metabolic markers of bone formation and resorption are also assessed in the Mayo Clinic patients.

Blood samples and mammographic, bone mineral density, and questionnaire data collected from patients randomized to receive exemestane on CAN-NCIC-MA27 are stored for future studies.

Patients complete a questionnaire at baseline, at 6-12 weeks, and at 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * Stage I, II, or III disease
  * Resected disease
* Planning to undergo treatment with anastrozole at the clinically approved dose of 1 mg/day OR Mayo Clinic Cancer Center Rochester patient who will be enrolled on or has been enrolled on CAN-NCIC-MA27 and has not started taking the study medication (anastrozole or exemestane)
* Hormone receptor status:

  * Estrogen receptor-positive and/or progesterone receptor-positive primary tumor

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal
* Able to complete questionnaires alone or with assistance

PRIOR CONCURRENT THERAPY:

* More than 6 months since prior endocrine therapy, except tamoxifen
* No other prior aromatase inhibitors (e.g., letrozole or exemestane)
* No prior ovarian function suppression with surgery or radiotherapy, ovarian ablation, or luteinizing hormone-releasing hormone analogues (e.g., goserelin) as treatment for cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of breast cancer. Stage I, II, or III disease.
  Planning to undergo treatment with anastrozole at the clinically approved dose of 1 mg/day OR Mayo Clinic Cancer Center Rochester patient who will be enrolled on or has been enrolled on CAN-NCIC-MA27 and has not started taking the study medication (anastrozole or exemestane)
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2005-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Association of single nucleotide polymorphisms with specific quantitative traits (i.e., hormone levels, breast density, and bone mineral density) | 4 years
Association of haplotype with traits | 4 years

SECONDARY OUTCOMES:
Association of genomic pathways with traits | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: James N. Ingle, MD, Principal Investigator — Mayo Clinic; Edith A. Perez, MD, Principal Investigator — Mayo Clinic; Donald W. Northfelt, MD, FACP, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas

REFERENCES:
- [Result] Ingle JN, Buzdar AU, Schaid DJ, Goetz MP, Batzler A, Robson ME, Northfelt DW, Olson JE, Perez EA, Desta Z, Weintraub RA, Williard CV, Flockhart DA, Weinshilboum RM. Variation in anastrozole metabolism and pharmacodynamics in women with early breast cancer. Cancer Res. 2010 Apr 15;70(8):3278-86. doi: 10.1158/0008-5472.CAN-09-3024. Epub 2010 Mar 30. PMID 20354183
- [Derived] Liu M, Goss PE, Ingle JN, Kubo M, Furukawa Y, Batzler A, Jenkins GD, Carlson EE, Nakamura Y, Schaid DJ, Chapman JA, Shepherd LE, Ellis MJ, Khosla S, Wang L, Weinshilboum RM. Aromatase inhibitor-associated bone fractures: a case-cohort GWAS and functional genomics. Mol Endocrinol. 2014 Oct;28(10):1740-51. doi: 10.1210/me.2014-1147. Epub 2014 Aug 22. PMID 25148458
- [Derived] Liu M, Ingle JN, Fridley BL, Buzdar AU, Robson ME, Kubo M, Wang L, Batzler A, Jenkins GD, Pietrzak TL, Carlson EE, Goetz MP, Northfelt DW, Perez EA, Williard CV, Schaid DJ, Nakamura Y, Weinshilboum RM. TSPYL5 SNPs: association with plasma estradiol concentrations and aromatase expression. Mol Endocrinol. 2013 Apr;27(4):657-70. doi: 10.1210/me.2012-1397. Epub 2013 Mar 21. PMID 23518928